CLINICAL TRIAL: NCT06024590
Title: Outcomes of Chlorhexidine Gluconate Irrigation as an Adjunctive Treatment in the Management of Diabetic Foot Ulcers
Brief Title: Outcomes of Irrisept Irrigation as an Adjunctive Treatment in the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Illinois Foot and Ankle Specialists (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIFAS-2023-001
Record Dates: First submitted 2023-08-28; First posted 2023-09-06 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A: irrigation with Irrisept™ (Active Comparator): Group A: standard of care wound treatment with 150 mL of IrriseptTM irrigation of the wound at each follow up visit.
  Interventions: Device: Irrisept
- Group B: irrigation or irrigation with normal saline (Active Comparator): Group B: standard of care wound treatment with 150 mL ration of normal saline irrigation of the wound at each follow up visit.
  Interventions: Device: Saline

INTERVENTIONS:
Device: Irrisept — Standard of care wound treatment with 150 mL of IrriseptTM irrigation of the wound at each follow up visit.
  Arms: Group A: irrigation with Irrisept™
Device: Saline — Standard of care wound treatment with 150 mL ration of Normal saline irrigation of the wound at each follow up visit
  Arms: Group B: irrigation or irrigation with normal saline

SUMMARY:
Irrisept™ irrigation containing Chlorhexidine Gluconate (CHG) 0.05% in sterile water, is an irrigation method that may help reduce bacterial load considerably more than traditional saline irrigation.

DETAILED DESCRIPTION:
The purpose of this clinical evaluation is to collect patient outcome data on Irrisept™ irrigation. This is a jet irrigation of 0.05% Chlorhexidine Gluconate (CHG) in sterile water delivered under pressure by manual compression of the bottle by the user. This treatment allows for management of bioburden in a wound through broad spectrum antimicrobial activity by the CHG as well as removal of debris from the wound bed.

In this trial, participants with partial and full thickness diabetic foot ulcers (DFUs) - 'full skin thickness and extending through the subcutaneous or fat layers or to deeper structures such as tendon and fascia will receive standard of care treatment with indicated off-loading device (SOC) for their condition in addition to wound bed irrigation with Irrisept™ or saline Irrigation.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Presence of a partial and full thickness DFU extending at least through the dermis and into the subcutaneous tissue down to the exposed tendon and fascia.
3. Wounds present anatomically on the foot as defined by beginning below the malleoli of the ankle, excluding wounds on the heel.
4. The index ulcer will be the largest ulcer if two or more eligible DFUs are present and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
5. Index ulcer (i.e., current episode of ulceration) has been present for greater than 4 weeks prior to first screening visit (SV1) and less than 1 year, as of the date the subject consents for study.
6. Adequate circulation to the affected foot as documented by the following: palpable pedal pulses, pulses audibly biphasic or triphasic with handheld doppler, or recent (<6 month) vascular testing (both invasive & non-invasive).
7. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
8. Subject understands and is willing to participate in the clinical study and can comply with weekly visits.
9. Subject understands they can exit the study at any time.

Exclusion Criteria:

1. Clinical signs of infection at the start of the study
2. Exposed bone(s)
3. Immunocompromised as determined by treating physician
4. Presence of greater than one full-thickness DFU less than 2 cm apart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the percentage of index ulcers healed at 12 weeks | Weekly up to 12 weeks
  Percentage of index ulcers healed from baseline up to 12 weeks

SECONDARY OUTCOMES:
Time: to heal within 12 weeks | Weekly up to 12 weeks
  Days to heal from baseline up to 12 weeks
Percent Area Reduction (PAR) at 12 weeks | Weekly up to 12 weeks
  Percent Area Reduction (PAR) from baseline up to 12 weeks
Pain reduction between visits, measured by Visual Analogue Scale (VAS) | Weekly up to 12 weeks
  Pain reduction from baseline up to 12 weeks. VAS (0-100 scale; 0 being no discomfort, 100 being intense discomfort)
Wound complication rate | Weekly up to 12 weeks
  Infection, return to operating room for management or other adverse events during the treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McEneaney, DPM, Principal Investigator — Northern Illinois Foot & Ankle Specialist
Locations (5):
- United States (5):
  - Northern Illinois Foot & Ankle Specialists, Cary, Illinois
  - Northern Illinois Foot & Ankle Specialists, Crystal Lake, Illinois
  - Northern Illinois Foot & Ankle Specialists, Elgin, Illinois
  - Northern Illinois Foot & Ankle Specialists, Fox Lake, Illinois
  - Northern Illinois Foot & Ankle Specialist, Lake in the Hills, Illinois

IPD SHARING:
Plan to Share IPD: No